CLINICAL TRIAL: NCT06019130
Title: Nivolumab in Combination With Cisplatin and 5-Fluorouracil as Induction Therapy in Children and Adults With EBV-positive Nasopharyngeal Carcinoma
Brief Title: Nivolumab in Children and Adults With Nasopharyngeal Carcinoma
Acronym: NPC-Nivo
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: German Society for Pediatric Oncology and Hematology GPOH gGmbH (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Principal Investigator, Prof. Dr. Udo Kontny, Head, Div. Pediatric Hematology, Oncology, Stem Cell Transplantation, RWTH Aachen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUCT: 2022-500676-59-00
Record Dates: First submitted 2023-08-15; First posted 2023-08-31 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Nasopharyngeal Carcinoma; Nasopharyngeal Cancer; Nasopharyngeal Neoplasms; Nasopharynx Cancer
Keywords: Immunotherapy; Nivolumab; Children; Adults; Chemotherapy; Immune Checkpoint Inhibitor
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Nasopharyngeal Neoplasms | interventions — Nivolumab; Cisplatin; Fluorouracil; Gemcitabine; Radiotherapy; Interferon beta-1a; Patient Reported Outcome Measures

STUDY DESIGN:
Intervention Model Description: A phase-II optimum Simon design with alpha=0.1 and beta=0.2 will be used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Patients < 26 years with non-metastatic disease with CR or PR after induction therapy (Experimental): Participants receive Nivolumab (4.5 mg/kg BW (max. 360 mg) every three weeks) during induction chemotherapy for a total of 3 doses, starting on day 1 of cycle 1 of induction standard chemotherapy with cisplatin 100 mg/m2 on day 1, plus 5-fluorouracil 1,000 mg/m2/d from day 1-5.
  After induction therapy patients will undergo standard radiochemotherapy. Primary PTV1 including elective irradiated LN-levels, will be 45Gy, with a boost ad 59.4Gy in patients with PR or a reduced boost at 54Gy in patients with CR. Cisplatin will be administered at 3x20mg/m2 in the first and last week of radiotherapy, each.
  Radiochemotherapy is followed by maintenance therapy with recombinant interferon-ß1a at 3x6Mio IU/week s.c. for 6 months.
  Interventions: Drug: Nivolumab; Drug: Cisplatin; Drug: 5-Fluorouracil; Radiation: Radiotherapy; Drug: Interferon beta-1a; Procedure: MRI; Procedure: PET; Behavioral: Patient-Reported Outcomes
- Patients < 26 y with no metastases and SD or PD after induction therapy or patients with metastases (Experimental): Participants receive Nivolumab (4.5 mg/kg BW (max. 360 mg) every three weeks) during induction chemotherapy for a total of 3 doses, starting on day 1 of cycle 1 of induction standard chemotherapy with cisplatin 100 mg/m2 on day 1, plus 5-fluorouracil 1,000 mg/m2/d from day 1-5. Patients with metastases responding to induction therapy may have a fourth cycle of induction therapy, including a fourth dose of Nivolumab.
  After induction therapy patients will undergo standard radiochemotherapy. Primary PTV1 including elective irradiated LN-levels, will be 45Gy, with a boost ad 59.4Gy. Cisplatin will be administered at 3x20mg/m2 in the first and last week of radiotherapy, each. Nivolumab (4.5 mg/kg BW (max. 360 mg) every three weeks) will be continued during radiochemotherapy, adding a total of 3 further doses of Nivolumab.
  Radiochemotherapy is followed by maintenance therapy with recombinant interferon-ß1a at 3x6Mio IU/week s.c. for 6 months.
  Interventions: Drug: Nivolumab; Drug: Cisplatin; Drug: 5-Fluorouracil; Radiation: Radiotherapy; Drug: Interferon beta-1a; Procedure: MRI; Procedure: PET; Behavioral: Patient-Reported Outcomes
- Patients >25 years with non-metastatic disease with CR or PR after induction therapy (Experimental): Participants receive Nivolumab (4.5 mg/kg BW (max. 360 mg) every three weeks) during induction chemotherapy for a total of 3 doses, starting on day 1 of cycle 1 of induction standard chemotherapy with cisplatin 100 mg/m2 on day 1, plus 5-fluorouracil 1,000 mg/m2/d from day 1-5.
  After induction therapy patients will undergo standard radiochemotherapy as outlined in current international guidelines (e.g. NCCN, ESMO).
  Interventions: Drug: Nivolumab; Drug: Cisplatin; Drug: 5-Fluorouracil; Radiation: Radiotherapy; Procedure: MRI; Procedure: PET; Behavioral: Patient-Reported Outcomes
- Patients > 25 years with non-metastatic disease with SD or PD after induction therapy (Experimental): Participants receive Nivolumab (4.5 mg/kg BW (max. 360 mg) every three weeks) during induction chemotherapy for a total of 3 doses, starting on day 1 of cycle 1 of induction standard chemotherapy with cisplatin 100 mg/m2 on day 1, plus 5-fluorouracil 1,000 mg/m2/d from day 1-5.
  After induction therapy patients will undergo standard radiochemotherapy as outlined in current international guidelines (e.g. NCCN, ESMO). Nivolumab (4.5 mg/kg BW (max. 360 mg) every three weeks) will be continued during radiochemotherapy, adding a total of 3 further doses of Nivolumab.
  Interventions: Drug: Nivolumab; Drug: Cisplatin; Drug: 5-Fluorouracil; Radiation: Radiotherapy; Procedure: MRI; Procedure: PET; Behavioral: Patient-Reported Outcomes
- Patients > 25 years with metastatic disease at diagnosis (Experimental): Participants receive Nivolumab (4.5 mg/kg BW (max. 360 mg) every three weeks) during induction chemotherapy for a total of 3 doses, starting on day 1 of cycle 1 of induction standard chemotherapy with cisplatin 80 mg/m2 on day 1, plus gemcitabine 1,000 mg/m2/d on day 1 and day 8, respectively. Patients responding to induction therapy may have a fourth cycle of induction therapy, including a fourth dose of Nivolumab.
  After induction therapy patients will undergo standard radiochemotherapy as outlined in current international guidelines (e.g. NCCN, ESMO). Nivolumab (4.5 mg/kg BW (max. 360 mg) every three weeks) will be continued during radiochemotherapy, adding a total of 3 further doses of Nivolumab.
  Interventions: Drug: Nivolumab; Drug: Cisplatin; Drug: Gemcitabine; Radiation: Radiotherapy; Procedure: MRI; Procedure: PET; Behavioral: Patient-Reported Outcomes

INTERVENTIONS:
Drug: Nivolumab — Nivolumab during induction chemotherapy in all groups and during radiochemotherapy in patients with SD or PD after induction or metastases
  Other Names: Opdivo
Drug: Cisplatin — Cisplatin during induction chemotherapy and during radiochemotherapy in all groups
  Other Names: Cisplatin Teva
Drug: 5-Fluorouracil — 5-Fluoruracil during induction chemotherapy in all groups except of adults > 25 years with metastatic disease at diagnosis
  Other Names: Fluorouracil-GRY
  Arms: Patients < 26 y with no metastases and SD or PD after induction therapy or patients with metastases; Patients < 26 years with non-metastatic disease with CR or PR after induction therapy; Patients > 25 years with non-metastatic disease with SD or PD after induction therapy; Patients >25 years with non-metastatic disease with CR or PR after induction therapy
Drug: Gemcitabine — Gemcitabine during induction chemotherapy in patients > 25 years with metastatic disease at diagnosis
  Other Names: Gemcitabin-GRY
  Arms: Patients > 25 years with metastatic disease at diagnosis
Radiation: Radiotherapy — After induction therapy in all patients
Drug: Interferon beta-1a — In patients < 26 years after end of radiochemotherapy for 6 months
  Other Names: Rebif
  Arms: Patients < 26 y with no metastases and SD or PD after induction therapy or patients with metastases; Patients < 26 years with non-metastatic disease with CR or PR after induction therapy
Procedure: MRI — At diagnosis and 17 to 22 days after the beginning of cycle 3 of induction therapy
Procedure: PET — At diagnosis and 17 to 22 days after the beginning of cycle 3 of induction therapy, either as PET-CT or PET-MRI
Behavioral: Patient-Reported Outcomes — For all patients at baseline, before radiochemotherapy, at day 100, and 2 years after enrolment

SUMMARY:
The purpose of this study is to assess whether the addition of the immune checkpoint inhibitor Nivolumab to induction chemotherapy will increase the percentage of patients with a complete response on MRI and PET after 3 cycles of induction therapy.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients will undergo a 2-week screening period to determine eligibility for study entry. After informed consent has been obtained, all patients ≤ 25 years and patients > 25 years without metastases will receive Nivolumab (4.5 mg/kg BW (max. 360 mg) q 3 weeks) added to standard induction chemotherapy (3 blocks of cisplatin/5-fluorouracil). In patients not responding to induction chemotherapy, the application of Nivolumab will be extended throughout the period of radiochemotherapy.

Patients > 25 years with metastatic disease will receive Nivolumab (4.5 mg/kg BW (max. 360 mg) q 3 weeks) added to induction chemotherapy with 3 blocks of cisplatin/gemcitabine.

All patients with metastatic disease will continue to receive Nivolumab during radiochemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed new diagnosis of nasopharyngeal carcinoma according to the current WHO classification in children and adolescents, aged between 3 years and 17 years, OR histologically confirmed new diagnosis of EBV-positive nasopharyngeal carcinoma, WHO stage II or III, in subjects ≥ 18 years
2. Stage II or higher in patients ≤ 25 years of age, stage III and IV in patients > 25 years of age (AJCC, 8th edition)
3. Measurable disease by MRI per RECIST 1.1 criteria
4. Sufficient tumor tissue to be sent for central review, including PD-L1 staining, either as 1 or 2 full blocks (preferred) or a minimum of 25 slides, obtained from core biopsy, punch biopsy, excisional biopsy or surgical specimen
5. Written informed consent by legal guardians (if patient not ≥ 18 years) and patient prior to study participation

Exclusion Criteria:

1. Newly diagnosed nasopharyngeal carcinoma, Stage I in all patients, Stage II in patients > 25 years of age
2. Recurrent nasopharyngeal carcinoma
3. Nasopharyngeal carcinoma diagnosed as second malignancy and preceding chemotherapy and/or radiotherapy
4. Prior chemotherapy and/or radiotherapy
5. Other active malignancy
6. Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
7. The subject received an investigational drug within 30 days prior to inclusion into this study
8. Subjects who are enrolled in another clinical trial
9. Subjects with prior organ allograft or allogenic bone marrow transplantation
10. Subjects with an active, known or suspected autoimmune disease. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enrol.
11. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days before start of therapy. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
12. Any positive test for hepatitis B virus or hepatitis C virus indicating acute or chronic infection
13. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
14. Inadequate hematologic, renal or hepatic function defined by any of the following screening laboratory values:

    1. WBC < 2 000/µl
    2. Neutrophils < 1 500/µl
    3. Platelets < 100 x 10e3/µL
    4. Hemoglobin < 9.0 g/dL
    5. Creatinine >1.5 x ULN or creatinine clearance < 50 mL/min (using the Cockcroft Gault formula or Schwartz formula in patients < 18 years)
    6. AST/ALT > 3 x ULN (> 5 x ULN if liver metastases)
    7. Total Bilirubin > 1.5 x ULN (except subjects with Gilbert Syndrome who must have a total bilirubin level ≥ 3.0 x ULN)
15. Hearing loss > 20 dB loss at 3 kHz due to an inner ear disorder and not caused by tumour burden
16. History of allergy or hypersensitivity to platinum-containing compounds or other study drug components
17. Clinically significant, uncontrolled heart disease (including history of any cardiac arrhythmias, e.g., ventricular, supraventricular, nodal arrhythmias, or conduction abnormality within 12 months of screening).
18. Vaccinated with live attenuated vaccines within 4 weeks of the first dose of the study drug.
19. Adequate performance status (Karnofsky score ≥ 60 for patients (age ≥ 16), Lansky score ≥ 60 (age < 16).
20. The subject has a history of any other illness, which, in the opinion of the Investigator, might pose an unacceptable risk by administering study medication.
21. The subject has any current or past medical condition and/or required medication to treat a condition that could affect the evaluation of the study.
22. Pregnant females as determined by positive [serum or urine] hCG test at Screening or prior to dosing. Participants of child-bearing age should use adequate contraception as defined in the study protocol. (Please refer to section 4.4)
23. Lactating females
24. Subjects, who are committed to an institution by virtue of an order issued either by the judicial or the administrative authorities
25. The subject is unwilling or unable to follow the procedures outlined in the protocol
26. The subject is mentally or legally incapacitated.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2026-01-09 (Estimated); Study Completion 2028-01-09 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate after induction therapy | MRI and PET will be done 17-22 days after start of induction therapy cycle 3 (each cycle is 21 days)
  Complete response by MRI and PET will be determined as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria

SECONDARY OUTCOMES:
Overall and Event-free Survival | 2 years after study enrolment
  Overall and event-free survival rates will be analysed with suitable descriptive methods (Kaplan Meyer estimates with confidence intervals) and compared with historical data using descriptive log-rank tests
Number of Treatment-Related Adverse Events | At day 0 of chemotherapy cycles 1, 2 and 3, each; at day 20-25 after beginning of chemotherapy cycle 3 (each cycle is 21 days); within 2-3 weeks after the last dose of radiotherapy; 100 days following the last dose of Nivolumab
  Adverse events will be classified using the National Cancer Institute Common Toxicity Criteria (NCI-CTCAE) version 5.0 by investigator assessment. Descriptive methods (frequency tables, rates of AE's and SAE's with 95% confidence intervals) will be applied
Efficacy based on PD-L1 expression in tumor tissue | Response to induction therapy will be measured 17-22 days after start of induction therapy cycle 3 (each cycle is 21 days), event-free and overall survival will be determined 2 years after study enrolment
  PD-L1-stained % of tumor cells at the time of diagnosis will be associated to the rate of response after induction therapy and EFS and OS

CONTACTS AND LOCATIONS:
Overall Officials: Udo Kontny, MD, Principal Investigator — Uniklinik RWTH Aachen
Locations (31):
- Germany (31):
  - Uniklinik RWTH Aachen, Department of Internal Medicine, Aachen
  - Uniklinik RWTH Aachen, Division of Pediatric Hematology, Oncology, Stem Cell Transplantation, Aachen
  - Department of Pediatric Oncology and Hematology, Charité University Medicine Berlin, Berlin
  - Evangelisches Klinikum Bethel, Children's Hospital, Bielefeld
  - Department of Pediatric Hematology and Oncology, University Hospital, Bonn
  - Department of Otorhinolaryngology, Head and Neck Surgery, University of Cologne, Cologne
  - Children's Hospital, Carl-Thiem Klinikum Cottbus, Cottbus
  - Clinic for Children and Adolescent Medicine, Klinikum Dortmund, Dortmund
  - Department of Internal Medicine, Klinikum Dortmund, Dortmund
  - Department of Pediatrics, University Hospital, Technische Universität Dresden, Dresden
  - Department fo Radiotherapy, University Hospital, Erlangen
  - Department of Pediatrics, University Hospital Erlangen, Erlangen
  - Department of Medical Oncology, West German Cancer Center, University Hospital Essen, Essen
  - Department of Pediatric Hematology and Oncology, University Hospital Essen, Essen
  - Department of Pediatrics, University Hospital, Frankfurt
  - Department of Pediatric Hematology/Oncology, University Hospital Freiburg, Freiburg im Breisgau
  - Department of Pediatric Oncology, Justus-Liebig University of Giessen, Giessen
  - Department of Pediatric Oncology, University Hospital, Göttingen
  - Department of Pediatric Hematology/Oncology, University Medicine Greifswald, Greifswald
  - Universitätsklinikum Halle, Klinik für Pädiatrie I, Halle
  - Department of Otorhinolaryngology, University Medical Center Hamburg-Eppendorf,, Hamburg
  - Department of Pediatric Oncology, University Children's Hospital, Hamburg
  - Department of Otorhinolaryngology, Jena University Hospital, Jena
  - Department of Pediatric Oncology, University Hospital Kiel, Kiel
  - Department of Pediatrics, University Hospital Mageburg, Magdeburg
  - Pediatric Hematology/Oncology, University Medicine Mainz, Mainz
  - Department of Otorhinolaryngology, Head and Neck Surgery, University Hospital Mannheim,, Mannheim
  - Department of Pediatric Hematology and Oncology, University Children's Hospital, Münster
  - Department of Pediatric Hematology, Oncology and Stem Cell Transplantation, University Hospital, Regensburg
  - Universitätsklinikum Tübingen, Klinik für Pädiatrie I, Tübingen
  - Department of Pediatric Hematology, Oncology and Stem Cell Transplantation, University Children's Hospital, University of Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No